CLINICAL TRIAL: NCT01426100
Title: A Randomized, Double-blind, Multi-center, Phase 3 Trial to Evaluate the Efficacy and Safety of a Fixed Dose Combination of Telmisartan and S-Amlodipine(CKD-828) Versus Telmisartan Monotherapy in Hypertensive Patients Inadequately Controlled by Telmisartan Monotherapy
Brief Title: CKD-828 Telmisartan Non-Responder Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 130HT11B
Record Dates: First submitted 2011-08-30; First posted 2011-08-31 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Hypertension
Keywords: CKD-828; Hypertension; Primary Hypertension; S-Amlodipine; Telmisartan; Amlodipine; Non-Responder
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — Telmisartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- CKD-828 40/2.5mg (Experimental)
  Interventions: Drug: CKD-828 40/2.5mg
- CKD-828 40/5mg (Experimental)
  Interventions: Drug: CKD-828 40/5mg
- Telmisartan 80mg (Active Comparator)
  Interventions: Drug: Telmisartan 80mg

INTERVENTIONS:
Drug: CKD-828 40/2.5mg — Fixed dose combination of Telmisartan 40mg and S-Amlodipine 2.5mg
  Arms: CKD-828 40/2.5mg
Drug: CKD-828 40/5mg — Fixed dose combination of Telmisartan 40mg and S-Amlidioine 5mg
  Arms: CKD-828 40/5mg
Drug: Telmisartan 80mg — Telmisartan 80mg monotherapy
  Arms: Telmisartan 80mg

SUMMARY:
The aim of the present study is to evaluate the efficacy and safety of two dose combination of Telmisartan/S-Amlodipine (40/2.5mg and 40/5mg) compared with telmisartan monotherapy (80mg) in hypertensive patients inadequately controlled by telmisartan monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* diagnosis of essential hypertension and blood pressure not adequately controlled(inadequate control defined as seated diastolic blood pressure(DBP)>= 90mmHg if on existing antihypertensive treatment of seated DBP >= 100mmHg if treatment naive)
* failure to respond to four weeks treatment with telmisartan 40mg(failure to respond defined as seated DBP >= 90mmHg)
* willing and able to provide written informed consent

Exclusion Criteria:

* mean seated DBP >= 120mmHg and/or mean seated SBP >= 200mmHg during run-in treatment or mean seated DBP >= 120mmHg and/or mean seated SBP >= 180mmHg at the randomization visit
* known or suspected secondary hypertension(ex. aortic coarctation, Primary hyperaldosteronism, renal artery stenosis, pheochromocytoma)
* has severe heart disease(Heart failure NYHA functional class 3, 4), unstable angina or myocardial infarction, arrhythmia within the past three months
* has cerebrovascular disease as cerebral infarction, cerebral hemorrhage within 6 months
* Type I Diabetes Mellitus, Type II Diabetes Mellitus with poor glucose control as defined by fasting glucosylated hemoglobin(HbA1c) > 8%
* nown severe or malignant retinopathy
* hepatic or renal dysfunction as defined by the following laboratory parameters: AST/ALT > UNL X 2, serum creatinine > UNL X 1.5
* acute or chronic inflammatory status need to treatment
* need to additional antihypertensive drugs during the study
* need to concomitant medications known to affect blood pressure during the study
* history of angioedema related to ACE inhibitors or Angiotensin II Receptor Blockers
* known hypersensitivity related to either study drug
* history of drug or alcohol dependency within 6 months
* any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of investigational products(ex. gastrointestinal tract surgery such as gastrectomy, gastroenterostomy or bypass, active inflammatory bowel syndrome within 12 months prior to screening, gastric ulcers need to treatment, gastrointestinal/rectal bleeding, impaired pancreatic function such as pancreatitis, obstructions of the urinary tract or difficulty in voiding
* administration of other study drugs within 30 days prior to randomization
* premenopausal women(last menstruation < 1year) not using adequate contraception, pregnant or breast-feeding
* history of malignancy including leukemia and lymphoma within the past 5 years
* in investigator's judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2011-08; Primary Completion 2012-05 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Mean Sitting Diastolic Blood Pressure (MSDBP) | After 8 weeks of treatment

SECONDARY OUTCOMES:
Mean Sitting Diastolic Blood Pressure (MSDBP) | After 4 weeks of treatment
Mean Sitting Systolic Blood Pressure (MSSBP) | After 4 weeks and 8 weeks of treatment
Response rate | After 4 weeks and 8 weeks of treatment
  Reduction of SBP ≥ 20mmHg, DBP ≥ 10mmHg
Control rate | After 4 weeks and 8 weeks of treatment
  Reduction SBP < 140mmHg, DBP < 90mmHg

CONTACTS AND LOCATIONS:
Locations (18):
- South Korea (18):
  - Kandong Sacred Heart Hospital, Anyang
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - DonGuk University Ilsan Hospital, Goyang
  - National Health Insurance Corporation Ilsan Hospital, Goyang
  - Gachon University Gil Medical Center, Inchon
  - Chonbuk National University Hospital, Jeonju
  - Seoul National University Bundang Hospital, Seongnam
  - Bundang Cha Medical Center, Seoul
  - Ewha Womans University Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Inje University Ilsan Paik Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyung Hee University Medical Center, Seoul
  - Severance Hospital, Seoul
  - Soon Chun Hyang University Hospital, Seoul
  - St. Paul's Hospital, The catholic University of Korea, Seoul
  - Ajou University Hospital, Suwon